CLINICAL TRIAL: NCT06540963
Title: Phase II Trial of Tipifarnib and Naxitamab for Relapsed/Refractory Neuroblastoma
Brief Title: Tipifarnib and Naxitamab for Relapsed/Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCC022
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — tipifarnib; naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HRNB Bone/Bone Marrow (Experimental): Cycles 1-6: Tipifarnib and Naxitamab Tipifarnib: on days 1-7 and 15-21 of each 28-day cycle. Naxitamab IV on Days 1, 3, and 5 of each cycle.
  Interventions: Drug: Tipifarnib; Drug: Naxitamab
- HRNB All others (Experimental): Cycles 1-6: Tipifarnib and Naxitamab Tipifarnib: on days 1-7 and 15-21 of each 28-day cycle. Naxitamab IV on Days 1, 3, and 5 of each cycle.
  Interventions: Drug: Tipifarnib; Drug: Naxitamab

INTERVENTIONS:
Drug: Tipifarnib — Tablet
  Other Names: R115777
Drug: Naxitamab — IV
  Other Names: Danyelza

SUMMARY:
The purpose of this study is to evaluate the investigational drug, tipifarnib (a pill taken by mouth), in combination with the Food and Drug Administration (FDA) approved drug, naxitimab, administered intravenously (IV; a liquid that continuously goes into your body through a tube that has been placed during a surgery into one of your veins). Naxitamab is FDA approved for pediatric patients 1 year of age and older and adult patients with relapsed or refractory high-risk neuroblastoma in the bone or bone marrow who have demonstrated a partial response, minor response, or stable disease to prior therapy, it may not be approved in the type of disease used in this study.

The goals of this part of the study are:

* Test the safety and tolerability of tipifarnib in combination with naxitimab in patients with cancer
* To determine the activity of study treatments chosen based on:
* How each subject responds to the study treatment
* How long a subject lives without their disease returning/progressing

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   Subjects must be age ≤ 21 years at initial diagnosis. Subjects must be >12 months of age at enrollment. Safety Run-In (first 6 subjects) must be age 6 years or older.
2. Pathology: All subjects must have a pathologically confirmed diagnosis of neuroblastoma at any point in their treatment.
3. Tumor assessment: Disease staging must be performed. This disease assessment is required for eligibility and must be done within a maximum of 4 weeks before first dose of study drug.
4. Disease Status: Relapsed/Refractory Neuroblastoma Relapsed disease defined as neuroblastoma that was previously in remission after standard therapy (at least 4 cycles of aggressive multi-drug induction chemotherapy, with or without radiation and surgery, followed by immunotherapy, or according to a standard high-risk treatment/neuroblastoma protocol) and has now relapsed and is in any number of relapses.

   Refractory disease defined as High-risk neuroblastoma as defined by the International Neuroblastoma Risk Group Staging System (INRG) that failed to achieve complete response (CR) after at least 4 cycles of aggressive multi-drug induction chemotherapy, progression during upfront therapy, or with disease remaining after standard immunotherapy.

   INRG High Risk NB defined as one of the following:
   1. Any age with International Neuroblastoma Risk Group (INRG) Stage L2, MS, or M with MYCN amplification
   2. Age ≥ 547 days and INRG Stage M regardless of biologic features
   3. Any age initially diagnosed with INRG Stage L1 MYCN amplified neuroblastoma (NBL) who have progressed to Stage M without systemic chemotherapy
   4. Age ≥ 547 days of age initially diagnosed with INRG Stage L1, L2, or MS who have progressed to Stage M without systemic chemotherapy
5. Measurable Disease: Subjects must be relapsed or refractory with active disease. Subjects must have measurable or evaluable disease, including at least one of the following: Measurable tumor >10mm by computed tomography scan (CT) or magnetic resonance imaging (MRI); a positive metaiodobenzylguanidine (MIBG) scan or positron emission tomography (PET) scan or Positive bone marrow biopsy/aspirate.
6. Subjects with central nervous system (CNS) disease currently taking steroids must have been on a stable dose of steroids for at least one week prior to their biopsy and must not have progressive hydrocephalus at enrollment.
7. Timing from prior therapy:

   Subjects must have fully recovered from the acute toxic effects of all prior anti- cancer chemotherapy and be within the following timelines:
   1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
   2. Hematopoietic growth factors: At least 5 days since the completion of therapy with a growth factor.
   3. Small Molecule Inhibitors (anti-neoplastic agent): At least 7 days since the completion of therapy with a small molecule inhibitor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
   4. Immunotherapy: At least 4 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines, CAR-T cells, anti-GD2 Monoclonal antibodies (ex. naxitamab, dinutuximab, etc.).
   5. XRT (Radiotherapy): At least 30 days since the last treatment except for radiation delivered with palliative intent to a non-target site.
   6. Stem Cell Transplant:

      * Allogeneic: No evidence of active graft vs. host disease
      * Allo/Auto: ≥ 2 months must have elapsed since transplant.
   7. MIBG Therapy: At least 6 weeks since treatment with MIBG therapy.
8. Subjects must have a Lansky or Karnofsky Performance Scale score of ≥ 50
9. Subjects must have adequate organ function at the time of enrollment:

   1. Hematological: Hematological recovery as defined by absolute neutrophil count (ANC) ≥750/μL, platelets ≥30/μL (may be transfused).
   2. Liver: Normal liver function as defined by Aspartate transferase (AST), Alanine transaminase (ALT), and total bilirubin (TBL) all within upper limit of normal
   3. Renal: Subjects must have adequate renal function defined as Creatinine clearance (in units ml/min) or radioisotope GFR ≥ 70. The formula to be used: Adjusted Glomerular Filtration Rate (GFR)=(Estimated GFR×BSA/1.73) mL/min.
   4. Cardiac: Subjects must have a QTcF ≤ 470 msc.
10. Subjects of childbearing potential must have a negative pregnancy test. Subjects of childbearing potential must agree to use an effective birth control method.
11. Subjects who are lactating must agree to stop breast-feeding. (NOTE: breast milk cannot be stored for future use while the mother is being treated on study.)
12. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or subjects' legal representative).

Exclusion Criteria:

1. Subjects who are less than 1 year of age
2. BSA of <0.25 m2
3. Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
4. Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
5. Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
6. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.
7. Previous Gr.4 allergic or anaphylactic reaction to naxitamab, leading to the discontinuation of naxitamab during prior therapy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the Overall Response Rate (ORR) of Participants using INSS Response | 6 months
  To evaluate the activity of Tipifarnib in combination with Naxitamab based on Overall response rate (ORR)

SECONDARY OUTCOMES:
Number of participants with progression free survival (PFS) during study | 6 months plus 5 years follow up
  To evaluate the activity of Tipifarnib in combination with Naxitamab based on Progression free survival (PFS)
Length of time that participants experience Overall Survival (OS) | 6 months plus 5 years follow up
  To evaluate the efficacy of Tipifarnib in combination with Naxitamab based upon Overall Survival (OS)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months plus 30 days
  To evaluate the safety and tolerability profile of Tipifarnib in combination with Naxitamab in pediatric and young adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Brown, MD, PhD, Study Chair — Beat Childhood Cancer
Locations (10):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Blood and Cancer Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Research Consortium website — https://research.beatcc.org/